CLINICAL TRIAL: NCT00001759
Title: Assessment of Lung Inflammation in Patients With Atopic Asthma Using Positron Emission Tomography
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980044; 98-I-0044
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Asthma; Hypersensitivity; Lung Diseases; Wegener's Granulomatosis
Keywords: Allergy; Fluorodeoxyglucose; Imaging; PET; Wegener's Granulomatosis; Asthma
MeSH Terms: conditions — Asthma; Hypersensitivity; Lung Diseases; Granulomatosis with Polyangiitis

SUMMARY:
Asthma is a chronic inflammatory disease. We propose to study inflammatory changes in the lungs of subjects with atopic asthma of different severity in vivo using positron emission tomography (PET) with 2-deoxy-2-[18F]fluoro-D-glucose (FDG). It has been shown that the uptake of FDG as detected by PET scanning correlates with inflammation in animal models as well as in human disease processes such as sarcoidosis, tuberculosis and abscess formation. In addition, it has been shown that the inflammation associated with allergen challenge in patients with atopic asthma can be visualized using PET scanning with FDG. We hypothesize that the degree of FDG-uptake as a measure of inflammation correlates with the severity of asthma as determined by pulmonary function tests and clinical signs and symptoms. In addition, information about the spatial distribution of the inflammatory changes will be obtained. To compare the characteristics of the inflammation in asthma with non-asthmatic inflammation of the lung, the images obtained in asthmatic subjects will be compared with images from subjects who have inflammatory changes of the lung caused by Wegener's granulomatosis. Subjects with atopic asthma and non-atopic control subjects will be selected from the community and, if eligible for the study, undergo skin testing against common allergens and pulmonary function testing. Subjects with Wegener's granulomatosis will be selected from a large group of subjects followed with this disease at NIAID. PET scanning with FDG will be used to measure inflammation in the PET scanning facility at the Clinical Center of the NIH and the results of the scanning will be correlated with the severity of the disease. We expect that for the first time this methodology will permit an objective measure of the basic pathogenic process, the allergic inflammation, in patients with atopic asthma. Using this methodology it will be possible to study the efficacy of currently available therapies for allergic inflammation. In addition, this methodology will provide an extremely useful tool for the development of new therapeutic approaches to the treatment of asthma.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disease. We propose to study inflammatory changes in the lungs of subjects with atopic asthma of different severity in vivo using positron emission tomography (PET) with 2-deoxy-2-[18F]fluoro-D-glucose (FDG). It has been shown that the uptake of FDG as detected by PET scanning correlates with inflammation in animal models as well as in human disease processes such as sarcoidosis, tuberculosis and abscess formation. In addition, it has been shown that the inflammation associated with allergen challenge in patients with atopic asthma can be visualized using PET scanning with FDG. We hypothesize that the degree of FDG-uptake as a measure of inflammation correlates with the severity of asthma as determined by pulmonary function tests and clinical signs and symptoms. In addition, information about the spatial distribution of the inflammatory changes will be obtained. To compare the characteristics of the inflammation in asthma with non-asthmatic inflammation of the lung, the images obtained in asthmatic subjects will be compared with images from subjects who have inflammatory changes of the lung caused by Wegener's granulomatosis. Subjects with atopic asthma and non-atopic control subjects will be selected from the community and, if eligible for the study, undergo skin testing against common allergens and pulmonary function testing. Subjects with Wegener's granulomatosis will be selected from a large group of subjects followed with this disease at NIAID. PET scanning with FDG will be used to measure inflammation in the PET scanning facility at the Clinical Center of the NIH and the results of the scanning will be correlated with the severity of the disease. We expect that for the first time this methodology will permit an objective measure of the basic pathogenic process, the allergic inflammation, in patients with atopic asthma. Using this methodology it will be possible to study the efficacy of currently available therapies for allergic inflammation. In addition, this methodology will provide an extremely useful tool for the development of new therapeutic approaches to the treatment of asthma.

ELIGIBILITY:
Subjects must be between 18 and 55 years of age.

Negative pregnancy test within two days of the scan and willingness to adhere to reliable birth control until the completion of the protocol.

Subjects must be able to give informed consent.

Subjects in the negative control group must have no history of asthma or other lung disease.

Control subjects must have negative prick skin tests to the allergens used.

Asthmatic subjects must have asthma as defined in this study.

Asthmatic subjects must have positive prick skin tests to one or more allergens used.

Subjects must have access to a primary medical care provider outside of the NIH.

Subjects must weigh less than 136 kg.

No breast feeding.

No smoking in the last 3 years, or greater than 6 months of smoking in the past ten years.

No antihistamines one week prior to the skin test on the first visit.

No history of coronary artery disease.

No evidence of lung disease other than asthma; no evidence of autoimmune or inflammatory disease which could affect lung function such as lupus erythematosus (except for the control subjects with Wegener's granulomatosis).

No evidence of either acute (e.g., bacterial or viral pneumonia) or chronic (e.g., bronchiectasis) lung infection.

No diabetes, or history of glucose intolerance (e.g., gestational diabetes).

No allergy to methacholine.

No beta-adrenergic blocking medication.

Control subjects must not have a history of asthma, atopic rhinitis or atopic dermatitis.

Control subjects must not have any response to inhaled methacholine with a fall in FEV1 in excess of 20% to less than or equal to 25 mg/ml.

Asthmatic subjects must not have chronic bronchitis or a diagnosis of chronic obstructive lung disease (COPD).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 95
Dates: Start 1997-12; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Floreani AA, Buchalter S, Thompson AB, Rennard SI. In vivo assessment of airway inflammation. Monaldi Arch Chest Dis. 1994 Jun;49(3 Suppl 1):17-26. PMID 8087134
- [Background] Taylor IK, Hill AA, Hayes M, Rhodes CG, O'Shaughnessy KM, O'Connor BJ, Jones HA, Hughes JM, Jones T, Pride NB, Fuller RW. Imaging allergen-invoked airway inflammation in atopic asthma with [18F]-fluorodeoxyglucose and positron emission tomography. Lancet. 1996 Apr 6;347(9006):937-40. doi: 10.1016/s0140-6736(96)91416-6. PMID 8598758
- [Background] Robinson DS, Hamid Q, Ying S, Tsicopoulos A, Barkans J, Bentley AM, Corrigan C, Durham SR, Kay AB. Predominant TH2-like bronchoalveolar T-lymphocyte population in atopic asthma. N Engl J Med. 1992 Jan 30;326(5):298-304. doi: 10.1056/NEJM199201303260504. PMID 1530827